CLINICAL TRIAL: NCT02381470
Title: Trial of Faropenem and Cefadroxil (in Combination With Amoxicillin/Clavulanic Acid and Standard TB Drugs) in Patients With Pulmonary Tuberculosis: Measurement of Early Bactericidal Activity and Effects on Novel Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faropenem_TB
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Tuberculosis
Keywords: Beta lactams; adjunctive therapy; drug-sensitive tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — fropenem; Amoxicillin-Potassium Clavulanate Combination; Cefadroxil; Rifampin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Faropenem (Experimental): Faropenem 600mg (with amoxicillin/clavulanic acid, 500mg/125mg) given three times daily for 7 days PLUS Rifampicin 10mg/kg once daily alone for the first 2 days then standard combination therapy (rifampicin, isoniazid, pyrazinamide, ethambutol, adjusted for body weight) for the following 5 days
  Interventions: Drug: Faropenem; Drug: Amoxicillin/clavulanic acid
- Cefadroxil (Experimental): Cefadroxil 1g (with amoxicillin/clavulanic acid, 500mg/125mg) given twice daily for 7 days PLUS Rifampicin 10mg/kg once daily alone for the first 2 days then standard combination therapy (rifampicin, isoniazid, pyrazinamide, ethambutol, adjusted for body weight) for the following 5 days
  Interventions: Drug: Amoxicillin/clavulanic acid; Drug: Cefadroxil
- Control (Active Comparator): Rifampicin 10mg/kg once daily alone for the first 2 days then standard combination therapy (rifampicin, isoniazid, pyrazinamide, ethambutol, adjusted for body weight) for the following 5 days
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Faropenem — Faropenem 600mg
  Other Names: Farobact 200
  Arms: Faropenem
Drug: Amoxicillin/clavulanic acid — Amoxicillin 500mg/ clavulanic acid 125mg
  Other Names: Augmentin; Co-amoxiclav
  Arms: Cefadroxil; Faropenem
Drug: Cefadroxil — Cefadroxil 1g
  Arms: Cefadroxil
Drug: Rifampicin — Rifampicin 10mg/kg
  Other Names: Rifampin
  Arms: Control

SUMMARY:
This trial aims to determine whether the early bactericidal activity of rifampicin given with faropenem or cefadroxil (each given with amoxicillin/clavulanic acid) is greater than the activity of rifampicin alone in patients with pulmonary TB. The trial will also investigate potential new biomarkers of sterilising activity.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the leading causes of mortality from an infectious disease worldwide with approximately 2 million deaths annually. There is an urgent need to identify new drugs, especially drugs with activity against persistent organisms that may enable shorter treatment regimens. Beta-lactam antibiotics have activity against TB in vitro and in animal models and there is evidence of synergy with rifampicin, one of the standard TB drugs. Amongst oral beta-lactam antibiotics, two appear to have optimal properties and optimal synergy with rifampicin and may be candidates for adjunctive treatment of drug-sensitive TB: faropenem (an oral penem, closely related to the carbapenem class) and cefadroxil (a first generation cephalosporin). Both drugs are used widely for the treatment of bacterial infections. They have in vitro activity against Mycobacterium tuberculosis, which is augmented when administered with rifampicin.

This is a Phase II randomised, controlled, open-label, early bactericidal activity trial. We will recruit patients between the ages of 18 and 70 with newly-diagnosed smear positive pulmonary TB, who have not yet started TB therapy.

Patients will be randomised into one of 3 arms to take faropenem (with amoxicillin/clavulanic acid) plus rifampicin, or cefadroxil (with amoxicillin/ clavulanic acid) plus rifampicin, or rifampicin alone for the first two days of the study. Patients will start standard TB therapy on the third day of the study and continue with the beta lactam antibiotics for the remaining 5 days of the study. Following the completion of the 7 days of study medication, the study will end and patients will continue standard combination TB therapy under normal clinical follow-up.

ELIGIBILITY:
Patient inclusion criteria:

1. Aged 18 to 70 years
2. Clinical features compatible with pulmonary TB
3. Sputum smear graded at least 1 +
4. Estimated to be producing at least 5ml of sputum per day
5. Willing to comply with study procedures and able to provide written informed consent.

Patient exclusion criteria:

1. Suspected miliary TB or TB meningitis
2. Patients receiving any TB treatment within the previous 6 months
3. Patients too ill to tolerate a 2-3 day delay in standard therapy
4. Concurrent bacterial pneumonia
5. Known hypersensitivity to beta-lactam drugs (penicillins, carbapenems) or rifampicin
6. History of severe allergies or severe asthma
7. Receiving loop diuretics
8. Estimated creatinine clearance < 80 ml/min on screening blood test
9. ALT > 2.5 times upper limit of normal on screening blood test.
10. Presence of rifampicin resistance on GeneXpert (or alternative molecular test).
11. Women who are currently pregnant or breastfeeding.
12. Any other significant condition that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial.
13. Participation in other clinical intervention trial or research protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Rate of change of time to positivity (TTP) in liquid culture from day 0 to day 2 | 2 days

SECONDARY OUTCOMES:
Rate of change of TTP in liquid culture from day 0 to day 7 | 7 days
Change in CFU/ml in solid culture from Day 0 to Day 2 | 2 days
Change in CFU/ml in solid culture from Day 0 to Day 7 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (6):
- Philippines (3):
  - De La Salle Health Institute, Cavite
  - Tropical Disease Foundation, Makati City
  - Lung Center Philippines, Quezon City
- National University Hospital, Singapore, Singapore, Singapore
- Uganda (2):
  - Infectious Diseases Institute, Kampala
  - Joint Clinical Research Centre, Kampala